CLINICAL TRIAL: NCT07235644
Title: Comparison of Efficacy and Safety in Patients Switching From MabThera® to Rixathon® in Relapsing-Remitting Multiple Sclerosis: an Observational Study
Brief Title: Comparison of Efficacy and Safety in Patients Switching From MabThera® to Rixathon® in Relapsing-Remitting Multiple Sclerosis
Status: Active, not recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-08358-01
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: MS (Multiple Sclerosis); Multiple Sclerosis (MS) - Relapsing-remitting; Multiple Sclerosis (Relapsing Remitting)
Keywords: Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Progressive Multiple Sclerosis; Rituximab; MabThera; Rixathon; Biosimilar; B-cell depletion; Neurofilament light chain (pNfL); MRI lesions; Disease progression; Disability progression; Expanded Disability Status Scale (EDSS); No Evidence of Disease Activity (NEDA); Quantitative MRI (qMRI); SyMRI; Plasma biomarkers; Observational Study; Retrospective Study; Treatment switch; Real-world evidence
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Charcot-Marie-Tooth disease, Type 1F; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS patients switched from MabThera® to Rixathon®: This cohort includes people with multiple sclerosis (MS) who were treated with MabThera® at Uppsala University Hospital and switched to Rixathon® starting January 2023 as part of routine clinical care. Participants were followed through standard clinical visits, blood tests, and MRI scans. Health outcomes before and after the switch will be compared using retrospective data from the Swedish MS Registry (SMSreg).

SUMMARY:
This observational study investigates if switching from MabThera® to Rixathon® is associated with changes in disease activity and/or safety in people with multiple sclerosis (MS).

The main questions it aims to answer are:

* Does switching to Rixathon® affect tissue damage, measured by blood levels of neurofilament light (pNfL)?
* Does switching to Rixathon® affect the number of new MRI lesions, relapses, or disability progression?

Researchers will look at health information already collected from participants before and after the medication switch. Participants include people with MS treated at Uppsala University Hospital who switched from MabThera® to Rixathon® starting in January 2023. Researchers will use data from regular clinical visits, blood tests, brain MRI scans, and disability scores (EDSS) recorded in the Swedish MS Registry.

DETAILED DESCRIPTION:
This is a retrospective observational study conducted at Uppsala University Hospital. The study aims to evaluate the efficacy and safety of switching from MabThera® (rituximab originator) to Rixathon® (rituximab biosimilar) in people with multiple sclerosis (MS), specifically those diagnosed with relapsing-remitting MS (RRMS) and progressive MS.

Starting in January 2023, the Department of Neurology at Uppsala University Hospital made an administrative decision to move from using rituximab (MabThera®) to rituximab (Rixathon®) in the treatment of MS, primarily for cost-saving reasons. This study will retrospectively analyze clinical and radiological outcomes collected before and after the switch. Data will be extracted from the Swedish MS Registry (SMSreg), a national database containing clinical information on people with MS across Sweden. Only patients treated at Uppsala University Hospital are included.

The primary objective of the study is to determine whether switching to Rixathon® affects disease activity, as measured by changes in plasma neurofilament light (pNfL) concentrations. pNfL is a biomarker of neuroaxonal damage, and elevated levels are associated with ongoing inflammation and neurodegeneration in MS.

Secondary objectives include comparing:

* The number of new T2 lesions on brain MRI scans before and after the switch
* The annualized relapse rate before and after the switch
* Changes in disability progression, measured by the Expanded Disability Status Scale (EDSS)
* Proportion of participants maintaining "No Evidence of Disease Activity" (NEDA) status
* Occurrence of serious adverse events (Grade 3-5 according to CTCAE v5.0)

Exploratory analyses will incorporate quantitative MRI (qMRI) metrics, including brain parenchymal fraction (BPF), myelin correlated fraction (MyCPF), myelin correlated volume (MyC), cerebrospinal fluid (CSF) volume, brain parenchymal volume (BPV), and intracranial volume. These parameters are obtained from SyMRI sequences that have been part of standard clinical practice at Uppsala University Hospital since 2017.

Participants eligible for inclusion were already being treated with MabThera® at the end of 2022 and completed the switch to Rixathon®. These individuals have been followed through routine clinical care with yearly MRI scans, regular EDSS assessments, and quarterly pNfL blood testing.

Data Quality Assurance:

Data will be obtained directly from SMSreg, which ensures quality through national standard operating procedures, regular audits, and predefined data validation rules. The registry will be vetted against clinical source documentation in the electronic medical records. Variables such as MRI findings, pNfL levels, relapse events, and EDSS scores are standardized across Sweden. No additional site-specific audits are planned beyond the SMSreg's internal quality controls.

Handling Missing Data:

In case of missing or inconsistent data points, standard imputation methods will be used as outlined in the analysis plan. For missing values that cannot be resolved, sensitivity analyses will be performed to assess the impact on results.

Sample Size and Power Considerations:

At the time of the medication switch, 184 MS patients were being treated with rituximab at the Department of Neurology. Given this sample size and historical relapse rates in RRMS, the study is adequately powered to detect meaningful differences in clinical and biomarker outcomes pre- and post-switch.

Statistical Analysis Plan:

The primary analysis will use a mixed-model repeated measures ANOVA to compare pNfL levels before and after the switch. Secondary outcomes (MRI activity, relapse rates, EDSS scores, NEDA status, and adverse events) will be analyzed using appropriate methods, including paired t-tests, Wilcoxon signed-rank tests, or McNemar's test, depending on the data distribution. Subgroup analyses will be performed separately for participants with RRMS and progressive MS. All analyses will adjust for potential confounders such as age, sex, disease duration, and prior treatment history.

This study will provide critical real-world evidence on whether switching to a rituximab biosimilar affects clinical outcomes and disease progression in MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple sclerosis (MS) according to the 2017 McDonald criteria (or previous applicable versions at the time of diagnosis).
* Treated with MabThera® (rituximab originator) at the Department of Neurology, Uppsala University Hospital before January 1, 2023.
* Switched to Rixathon® (rituximab biosimilar) for MS treatment starting January 1, 2023.
* Registered in the Swedish MS Registry (SMSreg) with available clinical data.
* At least one clinical follow-up visit recorded before the switch and one after the switch.
* Available plasma neurofilament light chain (pNfL) measurement and/or brain MRI scan during the study period.

Exclusion Criteria:

* No recorded clinical follow-up visit after switching to Rixathon®.
* Switched to Rixathon® but later discontinued treatment within 3 months for reasons unrelated to disease activity (e.g., administrative, insurance, or non-medical reasons).
* Participation in another interventional clinical trial affecting MS outcomes during the study period.
* Diagnosis of other major neurological diseases that could confound MS outcomes (e.g., stroke, CNS infection, or primary CNS tumors).
* Lack of consent for research use of data in the Swedish MS Registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected from people with multiple sclerosis (MS) treated at the Department of Neurology, Uppsala University Hospital, Sweden. All participants were registered in the Swedish MS Registry (SMSreg) and received MabThera® (rituximab originator) before switching to Rixathon® (rituximab biosimilar) as part of routine clinical care starting January 2023. The population includes individuals with relapsing-remitting MS and progressive MS who have available clinical follow-up data, blood biomarker measurements, and brain MRI scans.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in plasma neurofilament light chain (pNfL) levels before and after switching from MabThera® to Rixathon® | From the first available pNfL measurement (starting early 2022) to the time of data extraction in spring 2025
  Plasma neurofilament light chain (pNfL) is a blood biomarker that reflects nerve cell injury and disease activity in multiple sclerosis. Researchers will measure and compare pNfL levels collected before and after switching treatments to evaluate whether the switch influences underlying tissue damage. All available pNfL measurements from routine clinical practice will be used.

SECONDARY OUTCOMES:
Change in number of new T2 lesions on brain MRI before and after switching from MabThera® to Rixathon® | From earliest available MRI scans (starting in 2017) to the time of data extraction in spring 2025.
  Brain MRI scans will be used to assess new T2 lesions, a marker of disease activity in multiple sclerosis. Researchers will compare the number of new T2 lesions identified on MRI before and after switching treatments to evaluate the impact of the switch on radiological disease activity.
Change in annualized relapse rate before and after switching from MabThera® to Rixathon® | From earliest available clinical data (several years prior to 2023) to the time of data extraction in spring 2025.
  Relapse is defined as new or worsening neurological symptoms lasting at least 24 hours without external causes (such as fever or infection). Researchers will compare the annualized relapse rate before and after switching to assess the effect of the treatment change.
Change in disability progression measured by Expanded Disability Status Scale (EDSS) before and after switching from MabThera® to Rixathon® | From earliest available EDSS measurements (several years prior to 2023) to the time of data extraction in spring 2025.
  Disability progression will be evaluated using EDSS scores, a standardized method to quantify disability in MS. Researchers will compare EDSS scores to assess whether the treatment switch affects long-term disability progression.
Proportion of participants maintaining No Evidence of Disease Activity (NEDA) before and after switching from MabThera® to Rixathon® | From earliest available clinical and MRI data (several years prior to 2023) to the time of data extraction in spring 2025.
  NEDA is defined as absence of relapses, absence of new MRI lesions, and no confirmed disability worsening. Researchers will compare the proportion of participants maintaining NEDA status before and after the treatment switch.
Frequency of serious adverse events (Grade 3-5) after switching from MabThera® to Rixathon® | From the date of switching to Rixathon® (January 2023) to the time of data extraction in spring 2025.
  Serious adverse events will be recorded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Events graded 3-5 will be compared after the switch to evaluate safety outcomes associated with Rixathon® use.

OTHER OUTCOMES:
Change in quantitative MRI (qMRI) metrics using SyMRI before and after switching from MabThera® to Rixathon® | From earliest available SyMRI scans (starting in 2017) to the time of data extraction in spring 2025.
  Quantitative MRI (qMRI) metrics will be evaluated using SyMRI sequences collected during routine clinical care. Parameters assessed include brain parenchymal fraction (BPF), myelin correlated fraction (MyCPF), myelin correlated volume (MyC), cerebrospinal fluid (CSF) volume, brain parenchymal volume (BPV), and intracranial volume. Researchers will compare qMRI values before and after switching treatments to explore potential changes in brain structure and tissue integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Burman, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be made available upon request.
Supporting Information: Study Protocol, CSR
Time Frame: The data set will be stored for 15 years
Access Criteria: Study protocol will be made available upon request. Access to study data will be decided after contact with the study principal investigator. All access should be of scientific purposes.

REFERENCES:
- [Background] Simren J, Andreasson U, Gobom J, Suarez Calvet M, Borroni B, Gillberg C, Nyberg L, Ghidoni R, Fernell E, Johnson M, Depypere H, Hansson C, Jonsdottir IH, Zetterberg H, Blennow K. Establishment of reference values for plasma neurofilament light based on healthy individuals aged 5-90 years. Brain Commun. 2022 Jul 4;4(4):fcac174. doi: 10.1093/braincomms/fcac174. eCollection 2022. PMID 35865350
- [Background] McCamish M, Woollett G. The state of the art in the development of biosimilars. Clin Pharmacol Ther. 2012 Mar;91(3):405-17. doi: 10.1038/clpt.2011.343. Epub 2012 Feb 8. PMID 22318617
- [Background] Ventola CL. Biosimilars: part 1: proposed regulatory criteria for FDA approval. P T. 2013 May;38(5):270-87. PMID 23946620
- [Background] Calo-Fernandez B, Martinez-Hurtado JL. Biosimilars: company strategies to capture value from the biologics market. Pharmaceuticals (Basel). 2012 Dec 12;5(12):1393-408. doi: 10.3390/ph5121393. PMID 24281342
- [Background] Simoens S, Verbeken G, Huys I. Biosimilars and market access: a question of comparability and costs? Target Oncol. 2012 Dec;7(4):227-31. doi: 10.1007/s11523-011-0192-7. Epub 2012 Jan 17. PMID 22249657
- [Background] Hauser SL, Waubant E, Arnold DL, Vollmer T, Antel J, Fox RJ, Bar-Or A, Panzara M, Sarkar N, Agarwal S, Langer-Gould A, Smith CH; HERMES Trial Group. B-cell depletion with rituximab in relapsing-remitting multiple sclerosis. N Engl J Med. 2008 Feb 14;358(7):676-88. doi: 10.1056/NEJMoa0706383. PMID 18272891
- [Background] Svenningsson A, Frisell T, Burman J, Salzer J, Fink K, Hallberg S, Hambraeus J, Axelsson M, Nimer FA, Sundstrom P, Gunnarsson M, Johansson R, Mellergard J, Rosenstein I, Ayad A, Sjoblom I, Risedal A, de Flon P, Gilland E, Lindeberg J, Shawket F, Piehl F, Lycke J. Safety and efficacy of rituximab versus dimethyl fumarate in patients with relapsing-remitting multiple sclerosis or clinically isolated syndrome in Sweden: a rater-blinded, phase 3, randomised controlled trial. Lancet Neurol. 2022 Aug;21(8):693-703. doi: 10.1016/S1474-4422(22)00209-5. PMID 35841908
- [Background] Brown JWL, Coles A, Horakova D, Havrdova E, Izquierdo G, Prat A, Girard M, Duquette P, Trojano M, Lugaresi A, Bergamaschi R, Grammond P, Alroughani R, Hupperts R, McCombe P, Van Pesch V, Sola P, Ferraro D, Grand'Maison F, Terzi M, Lechner-Scott J, Flechter S, Slee M, Shaygannejad V, Pucci E, Granella F, Jokubaitis V, Willis M, Rice C, Scolding N, Wilkins A, Pearson OR, Ziemssen T, Hutchinson M, Harding K, Jones J, McGuigan C, Butzkueven H, Kalincik T, Robertson N; MSBase Study Group. Association of Initial Disease-Modifying Therapy With Later Conversion to Secondary Progressive Multiple Sclerosis. JAMA. 2019 Jan 15;321(2):175-187. doi: 10.1001/jama.2018.20588. PMID 30644981
- [Background] Lizak N, Lugaresi A, Alroughani R, Lechner-Scott J, Slee M, Havrdova E, Horakova D, Trojano M, Izquierdo G, Duquette P, Girard M, Prat A, Grammond P, Hupperts R, Grand'Maison F, Sola P, Pucci E, Bergamaschi R, Oreja-Guevara C, Van Pesch V, Ramo C, Spitaleri D, Iuliano G, Boz C, Granella F, Olascoaga J, Verheul F, Rozsa C, Cristiano E, Flechter S, Hodgkinson S, Amato MP, Deri N, Jokubaitis V, Spelman T, Butzkueven H, Kalincik T; MSBase Study Group. Highly active immunomodulatory therapy ameliorates accumulation of disability in moderately advanced and advanced multiple sclerosis. J Neurol Neurosurg Psychiatry. 2017 Mar;88(3):196-203. doi: 10.1136/jnnp-2016-313976. Epub 2016 Sep 28. PMID 27683916
- [Background] Capra R, Cordioli C, Rasia S, Gallo F, Signori A, Sormani MP. Assessing long-term prognosis improvement as a consequence of treatment pattern changes in MS. Mult Scler. 2017 Nov;23(13):1757-1761. doi: 10.1177/1352458516687402. Epub 2017 Jan 12. PMID 28080255